CLINICAL TRIAL: NCT03527290
Title: Dietary Approaches for Improving Cardiometabolic Health
Brief Title: Dietary Approaches for Cardiometabolic Health
Acronym: DACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Andrew Odegaard, Assistant Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-3929
Record Dates: First submitted 2018-04-26; First posted 2018-05-17 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Abdominal; Dyslipidemias; Insulin Resistance; Blood Pressure; Weight Loss
MeSH Terms: conditions — Obesity, Abdominal; Dyslipidemias; Insulin Resistance; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants are blinded to the nature of the other intervention so as not to contaminate the intervention. The clinical research staff taking the measurements is also blinded to the respective intervention the participant has been randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (Experimental): Participants will be instructed and counseled to incorporate a 12-hour Time Restricted Eating (TRE) regimen that begins upon waking and concludes within a 12-hour period (e.g. if wake at 6:30 AM then all caloric intake occurs between 6:30 AM and 6:30 PM). Water and non-caloric beverages (e.g. herbal tea) outside the period are encouraged as desired. There are no specific content or energy intake changes to the diet counseled or recommended as the focus of the counseling in this arm is timing of eating with innate circadian patterns and developing plans and approaches to follow this plan.
  Interventions: Behavioral: Time Restricted Eating
- Standard Cardiometabolic Health Diet (Active Comparator): Participants will be instructed and counseled with standard clinical dietary guidance for improving cardiometabolic health, where the focus is on the content, specifically a dietary pattern that emphasizes vegetables, fruits, whole grains, legumes, nuts/seeds, low fat dairy, seafood, lean poultry and meat and avoidance of foods with high levels of sodium, added sugars, saturated fats, and trans fats. There is no prescription to reduce energy intake.
  Interventions: Behavioral: Standard Cardiometabolic Health Diet

INTERVENTIONS:
Behavioral: Time Restricted Eating — The intervention is delivered in a paradigm in which an individual with abdominal obesity would be referred by their physician to receive dietary counseling from a Registered Dietitian (RD). The aim of the intervention is to improve cardiometabolic health and assist with weight management via 4, individualized counseling sessions over the course of 8 weeks. Participants are educated on basic concepts related to circadian rhythms, metabolism and TRE; and the evidence demonstrating benefit of TRE in animal models and humans. The goal is provide rationale for the potential benefits of a TRE approach. In addition, the RD sessions focus on developing a plan for successfully implementing a TRE approach, identifying challenges for adherence, and a plan for dealing with real or potential challenges. The counseling is focused the TRE concept, with no specific direction or counseling related to modifying the content of the participant's diet or any prescription to reduce energy intake.
  Other Names: TRE
  Arms: Time Restricted Eating
Behavioral: Standard Cardiometabolic Health Diet — The intervention is delivered in a paradigm in which an individual with abdominal obesity would be referred by their physician to receive dietary counseling from a Registered Dietitian (RD). The aim of the intervention is to improve cardiometabolic health and assist with weight management via 4, individualized counseling sessions over the course of 8 weeks. Participants are educated on basic concepts and known benefits related to eating a diet for cardiometabolic health and weight management recommended by the American Heart Association and the Academy of Nutrition and Dietetics as a standard of practice for dietitians in healthcare settings. The RD sessions focus on adopting a dietary pattern aligned with this approach, identifying challenges to adopting this dietary pattern, and education and plans for dealing with real or potential challenges. The counseling gives no direction related to modifying the timing of dietary intake or any prescription to reduce energy intake.
  Other Names: STD
  Arms: Standard Cardiometabolic Health Diet

SUMMARY:
This pilot study aims to recruit 30 adults with abdominal obesity, without major chronic disease, and test whether clinical dietary advice that is solely focused on the timing of eating (time restricted eating), has an effect on cardiometabolic health compared to standard dietary advice for cardiometabolic health, which is focused on content. The goal of this pilot study is to develop and hone dietary counseling approaches for time restricted eating for RD's in a clinical practice paradigm, and collect data on testing this intervention compared to standard dietary counseling approaches for cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal obesity (waist circumference ≥35" for women and ≥40" for men; if Asian ethnicity, ≥35" for men and ≥31.5" for women)
* weight stable over the previous 2 months
* medications stable for > 3 months
* self-reported 24-hr sleep-wake patterns within the appropriate range as defined by the National Sleep Foundation (self-reported habitual sleep duration 6-10 hours during nocturnal hours)
* regular meal patterns
* from the greater UCI and Orange county area
* willing to incorporate a dietary approach aimed at improving cardiometabolic health and weight management
* able to speak, read and understand English or Spanish

Exclusion Criteria:

* Self-reported unstable hypertension
* Type 1 or 2 diabetes mellitus
* heart, renal, or liver disease
* cancer or active neoplasms
* hyperthyroidism unless treated and under control
* taking any medications known to affect clinical risk measures of interest or weight/energy expenditure (except for stable blood pressure medication)
* active usual smoking (tobacco or marijuana)
* alcohol intake > 3 drinks/day
* pregnancy, current lactation, or plans to become pregnant during the study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Triglyceride : HDL cholesterol ratio | 8 weeks
  Ratio of fasting triglycerides to HDL cholesterol

SECONDARY OUTCOMES:
HOMA-IR | 8 weeks
  Estimation of HOMA-IR from fasting glucose and insulin
Glucose | 8 weeks
  Fasting glucose
Insulin | 8 weeks
  Fasting insulin
LDL cholesterol | 8 weeks
  LDL cholesterol
Weight | 8 weeks
  Body weight measured on calibrated scale
Waist Circumference | 8 weeks
  Measured by standard approach utilized in NHANES
Diet Quality | Run-in (up to 2 weeks), Intervention (8 weeks)
  Assessed by 2 unannounced recalls during run-in period and 3 during intervention
Post-hoc estimated energy intake | 8 weeks
  Estimated by utilizing NIDDK Body weight planner with weights measured over 8 weeks
Objective sleep and physical activity habits | Run-in (up to 2 weeks), Intervention (8 weeks)
  Measured with fitbit
Blood pressure | 8 weeks
  Resting systolic and diastolic blood pressure

OTHER OUTCOMES:
Eating duration | Run-in (up to 2 weeks), Intervention (8 weeks)
  Glycemic data from blinded continuous glucose monitor to estimate actual daily eating period

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Odegaard, PhD, MPH, Principal Investigator — University of California, Irvine
Locations (1):
- Institute for Clinical and Translational Science, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to make this available to other researchers upon completion of the pilot study, publication, and receiving IRB approval to do so.